CLINICAL TRIAL: NCT03795857
Title: Lethal Fetal Abnormality : the Experience of Pregnancy by Parents Who Have Chosen to Carry to Term With Palliative Care.
Brief Title: Antenatal Palliative Care
Acronym: SPAN
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0371
Record Dates: First submitted 2019-01-02; First posted 2019-01-08 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Fetal Death; Fetal Anomaly
MeSH Terms: conditions — Fetal Death; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Semi-structured interviews — The purpose of this study is to describe the experience of pregnancy by parents who have chosen to carry to term despite a lethal fetal diagnosis. Therefore, semi-structured interviews will be conducted to explore the links between context, feeling, involvement, decision and actions during pregnancy, whether within the couple or in its environment.

SUMMARY:
In France, according to current legislation, termination of pregnancy could be performed without any upper gestational age limit, if there is a strong probability that the fetus will be affected by a particularly severe and incurable disease. When there is a lethal fetal diagnosis most of parents wish to terminate their pregnancy. However, and despite some medical resistance a few of them do wish to continue pregnancy. In these situations, palliative care seems to be a good way to prepare to welcome the child and surround him until death.

The aim of the study is to describe parents' experience for a better understanding and a better care.

ELIGIBILITY:
Inclusion Criteria:

* The woman must be between the ages of 18 and 50 and the adult,
* Participants must have received the information and not have objected to participating in the study,
* the lethal / adverse short-term prognosis of the fetal pathology must have been confirmed by a committee of experts (CPDPN),
* The choice to continue the pregnancy should have been clearly expressed,
* The birth of the child should not be older than 24 months.
* The child's death must be more than 6 months old (or not have occurred)

Exclusion Criteria:

* Non-mastery of the French language,
* Measure of legal protection of one of the members of the couple (guardianship, trusteeship, ...),
* Severe psychiatric or neurological disorders inducing significant cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will focus on couples who have been diagnosed with lethal fetal pathology and who have chosen to continue the pregnancy for a birth in palliative care.
  The death of the child may have occurred in utero or after birth.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Description of the pregnancy by parents who have chosen to carry to term despite a lethal fetal diagnosis | About 1 hour and 30 minutes
  The purpose of this study is to describe the experience of pregnancy by parents who have chosen to carry to term despite a lethal fetal diagnosis. Therefore, semi-structured interviews will be conducted to explore the links between context, feeling, involvement, decision and actions during pregnancy, whether within the couple or in its environment.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Équipe de psychopathologie périnatale - Service de psychopathologie du développement - Centre Hospitalier Femme-Mère-Enfant - Hospices Civils de Lyon, Bron
  - Service de gynécologie obstétrique - Hôpital de la Croix Rousse, Lyon
  - Service de gynécologie-obstétrique - Centre hospitalier Lyon sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No